CLINICAL TRIAL: NCT03924635
Title: A 24-week Randomised Exploratory Open-Label Study Aiming To Characterise Changes In Airway Inflammation, Symptoms, Lung Function, And Reliever Use In Asthma Patients Using SABA (Salbutamol) Or Anti-Inflammatory Reliever (SYMBICORT®) As Rescue Medication In Addition To SYMBICORT As Daily Asthma Controller
Brief Title: An Exploratory Study to Characterise Changes in Airway Inflammation, Symptoms, Lung Function and Reliever Use in Adult Asthma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D589BC00018; 2018-003467-64 (EudraCT Number)
Record Dates: First submitted 2019-01-31; First posted 2019-04-23 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Airway Inflammation; Asthma
Keywords: Airway inflammation; Anti-inflammatory reliever; SYMBICORT; Maintenance anti-inflammatory therapy; Reliever medication; Salbutamol
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Albuterol; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SYMBICORT as maintenance and reliever treatment (Active Comparator): Patients on ICS (low dose)/LABA prior to study entry will receive SYMBICORT (budesonide/formoterol 100/6 μg) × 2 twice a day (BID) for maintenance and as needed (PRN) for relief and patients on ICS (medium dose)/LABA prior to study entry will receive SYMBICORT (budesonide/formoterol 200/6 μg) × 2 BID for maintenance and PRN for relief.
  Interventions: Combination Product: SYMBICORT and salbutamol
- SYMBICORT as maintenance, salbutamol as reliever treatment (Active Comparator): Patients on ICS (low dose)/LABA prior to study entry will receive SYMBICORT (budesonide/formoterol 100/6 μg) × 2 BID for maintenance + salbutamol (100 μg) PRN for relief and patients on ICS (medium dose)/LABA prior to study entry will receive SYMBICORT (budesonide/formoterol 200/6 μg) × 2 BID for maintenance + salbutamol (100 μg) PRN for relief.
  Interventions: Combination Product: SYMBICORT and salbutamol

INTERVENTIONS:
Combination Product: SYMBICORT and salbutamol — SYMBICORT will be given in a TURBOHALER. Salbutamol will be given in a pressurised metered dose inhaler.
  Other Names: VENTOLIN (salbutamol); SYMBICORT (budesonide/formoterol)

SUMMARY:
This is a randomised, active-comparator, open-label, parallel-group, multicentre phase IV exploratory study to characterise changes in airway inflammation, symptoms, lung function, and reliever use in asthma patients using SABA (salbutamol) or anti inflammatory reliever (SYMBICORT®) as reliever medication in addition to SYMBICORT as daily asthma controller. Eligible patients diagnosed with asthma at least 6 months prior to the Screening Visit (Visit 1) and fulfilling all of the inclusion criteria and none of the exclusion criteria will continue into the Run-in Period. At Visit 2, patients will be assessed for randomisation criteria and, if met, will be randomised to receive either SYMBICORT as maintenance and reliever treatment or SYMBICORT as maintenance treatment and salbutamol as reliever treatment in a 1:1 ratio. Randomisation will be stratified by the patient's ongoing dose of inhaled corticosteroids [(ICS) low or medium] at study entry

DETAILED DESCRIPTION:
This is a randomised, active-comparator, open-label, parallel-group, multicentre phase IV exploratory study to characterise changes in airway inflammation, symptoms, lung function, and reliever use in asthma patients using SABA (salbutamol) or anti-inflammatory reliever (SYMBICORT®) as reliever medication in addition to SYMBICORT as daily asthma controller. Eligible patients diagnosed with asthma at least 6 months prior to the Screening Visit (Visit 1) and fulfilling all of the inclusion criteria and none of the exclusion criteria will continue into the Run-in Period. During the run-in period, patients will take their maintenance medication (ie, SYMBICORT [100/6 or 200/6 μg, × 2 BID]) and reliever salbutamol [100 μg, PRN]) using the connected inhalers. At Visit 2, patients will be assessed for randomisation criteria and, if met, will be randomised to receive either SYMBICORT as maintenance and reliever treatment or SYMBICORT as maintenance treatment and salbutamol as reliever treatment in a 1:1 ratio. Randomisation will be stratified by the patient's ongoing dose of ICS (low or medium) at study entry. This study will include a minimum of 3 site visits. Patients will be requested to come to the study site for 4 additional Event Visits (E1 to E4) at approximately 4-day intervals beginning after the first visit if they experience any one of the following 3 criteria: a) A severe exacerbation defined as use of systemic steroids for at least 3 days, emergency room visit, or inpatient hospitalisation due to asthma, b) Symptom worsening criteria based on CompEx evaluation - an asthma worsening identified by a combination of deteriorations in at least 2 variables (decrease in PEF of at least 15% compared with baseline, an increase of reliever medication of at least 1.5 occasions compared with baseline, or an increase in asthma symptoms of at least 1 compare with baseline or the absolute max score [=3]) at least 2 consecutive days, or c) A single day (in 24 hours) with 6 or more occasions of reliever medication use.

The duration of participation in the study will be 26 to 28 weeks (maximum) for each individual patient, including a 2-week Run-in Period, followed by a 24-week randomised Treatment Period and an additional follow-up period if the Event Visits fall within the final 2 weeks of the Treatment Period. The study plans to randomise a minimum of 60 patients to a maximum of 80 patients to achieve at least 54 patients completing the study. The study will be conducted at no less than 2 sites in the United Kingdom (UK). The estimated study duration is approximately 30 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written Informed Consent Form (ICF) prior to any study-related procedures, sampling, and analyses (at Visit 1).
2. Patient must be ≥18 years of age at the time of signing the ICF.
3. A physician diagnosis of asthma for a minimum ≥6 months prior to Visit 1.
4. Use of ICS (low or medium dose)/LABA for asthma for ≥3 months prior to Visit 1.
5. Episode of asthma symptom worsening requiring overuse of reliever (more than the standard for the individual patient) at least once during the last 30 days prior to Visit 1.
6. The patient must be able to read speak, and understand local language; and be able to, in the Investigator's judgment, comply with the study protocol.
7. Able to perform home FeNO and spirometry assessments and complete the asthma symptom diary on a regular basis during the conduct of the study.
8. Male and/or female
9. Negative pregnancy test (urine) for female patients of childbearing potential at Visit 1.
10. For randomisation at Visit 2, patients should fulfil the following criteria:

    1. Symptoms requiring reliever medication use for a minimum of 2 to a maximum 8 days out of the last 10 days of the Run-in Period.
    2. At least 80% overall compliance rate for performing FeNO and spirometry assessments and completing the asthma symptom diary during the Run-in Period.

Exclusion Criteria:

1. Any significant disease or disorder, or evidence of drug/substance abuse which in the Investigator's opinion would pose a risk to patient safety, interfere with the conduct of study, have an impact on the study results, or make it undesirable for the patient to participate in the study.
2. Any asthma worsening requiring change in asthma treatment other than the patient's prescribed reliever medication (SYMBICORT as Maintenance and Reliever Therapy [SMART] therapy, SABA, and/or short-acting anticholinergic agent) within 30 days prior to Visit 1.
3. Medical history of life- threatening asthma including intubation and intensive care unit admission.
4. Medical conditions (other than allergic rhinitis) or medications (other than ICS) that will influence FeNO, as judged by the Investigator.
5. Concurrent respiratory disease: presence of a known pre-existing, clinically important lung condition other than asthma (eg, cystic fibrosis, idiopathic pulmonary fibrosis, pulmonary arterial hypertension).
6. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained (Visit 1) or during the screening/Run-in Period.
7. A severe asthma exacerbation (defined by an exacerbation resulting in ≥3 days of oral corticosteroids [or one depot intramuscular injection of a glucocorticosteroid], an urgent care or emergency room visit that results in systemic corticosteroids, or an inpatient hospitalisation due to asthma) within 30 days prior to screening.
8. Any disease state or procedure that may necessitate the use of oral/systemic corticosteroids during the Treatment Period, other than asthma.
9. Malignancy: a current malignancy or previous history of cancer in remission for less than 12 months prior to Visit 1 (patients that had localised carcinoma of the skin which was resected for cure will not be excluded).
10. Patients with a history/treatment of malignancy, and which in the Investigator's opinion could compromise the safety of the patient.
11. Other concurrent medical conditions: patients who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
12. Current smokers: previous smokers are allowed to be included provided that they stopped smoking >12 months prior to Visit 1 AND have a smoking history of ≤10 pack-years.
13. Alcohol/substance abuse: a history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.
14. Participation in another clinical study with any marketed or investigational biologic drug within 4 months or 5 half-lives (whichever is longer) prior to Visit 1.
15. Participation in another clinical study with a non-biologic investigational product or new formulation of a marketed non-biologic drug during the last 30 days prior to Visit 1.
16. Patients with a known hypersensitivity to the study drugs or any of the excipients of the products.
17. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
18. Previous randomisation in the present study.
19. For women only: currently pregnant (confirmed with positive pregnancy test), breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the Investigator. Periodic abstinence, spermicides only, and the lactational amenorrhoea method are not acceptable methods of contraception.
20. Planned hospitalisation during the study that would interfere with study objectives as judged by the Investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Research Site, Bradford
  - Research Site, Dundee
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Watford
  - Research Site, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BC00018&attachmentIdentifier=8fc1d44e-d319-4346-966a-1e1338372603&fileName=D589BC00018_(PXL_241309)_Redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at six study sites in United Kingdom between 01 August 2019 and 16 December 2022.
Pre-assignment Details: Eligible patients from the screening visit entered the 14-day run-in period during which they used 4 devices (1 spirometry sensor, 1 FeNO device, and 2 inhaler sensors) connected to the STIFLE App. The Investigator (or trained study staff) ensured all devices were connected properly and instructed patients on how to use each device and the STIFLE App prior to the run-in period.
Groups:
- SYMBICORT as Maintenance and Reliever Treatment: Patients on ICS (low dose)/LABA prior to study entry received SYMBICORT (budesonide/formoterol 100/6 μg) × 2 twice a day (BID) for maintenance and as needed (PRN) for relief and patients on ICS (medium dose)/LABA prior to study entry received SYMBICORT (budesonide/formoterol 200/6 μg) × 2 BID for maintenance and PRN for relief.
- SYMBICORT as Maintenance, Salbutamol as Reliever Treatment: Patients on ICS (low dose)/LABA prior to study entry received SYMBICORT (budesonide/formoterol 100/6 μg) × 2 BID for maintenance + salbutamol (100 μg) PRN for relief and patients on ICS (medium dose)/LABA prior to study entry received SYMBICORT (budesonide/formoterol 200/6 μg) × 2 BID for maintenance + salbutamol (100 μg) PRN for relief.
Period: Overall Study
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Started | 18 | 24
Completed | 16 | 20
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all patients randomised who had at least 1 post baseline measurement, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment | Total
Number analyzed (Participants) | 18 | 24 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (14.6) | 45.5 (16.0) | 49.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 0 | 0 | 0
  Race: White | 17 | 22 | 39
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 0 | 0 | 0
  Race: Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO was measured by the patient using a FeNO monitoring device (Vivatmo Me). Standard deviation of daily measurement of FeNO were presented for each patient and based on these summary statistics at treatment level were calculated.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: The FAS was defined as all patients randomised who had at least 1 post baseline measurement, irrespective of their protocol adherence and continued participation in the study.
Measure: Mean (Full Range); unit: parts per billion (ppb)
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
parts per billion (ppb) | 8.67 [3.25 to 23.97] | 9.01 [2.28 to 18.58]

2. Primary Outcome: Total Asthma Symptoms Score
Description: Symptoms scores were calculated using the asthma symptom diary.
  Asthma symptoms during daytime and night-time were recorded by the patient twice daily in the asthma symptom diary, according to the following scoring system:
  0 = no asthma symptoms
  1. = you are aware of your asthma symptoms, but you can easily tolerate the symptoms
  2. = your asthma is causing you enough discomfort to cause problems with normal activities (or with sleep)
  3. = you are unable to do your normal activities (or to sleep) because of your asthma
  Total asthma symptom scores were reported, which were calculated as the sum of non-missing morning and evening scores. Lower scores indicate no impairment/symptoms, representing increased asthma control. Conversely, higher scores indicate more severe impairment/symptoms, indicating reduced asthma control.
  Standard deviation of total (daily) asthma symptom scores were presented for each patient and based on these summary statistics at treatment level were calculated.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Score on a scale | 0.58 [0.08 to 1.26] | 0.83 [0.00 to 1.47]

3. Primary Outcome: Total Reliever Medication Use
Description: Reliever medication usage was captured in the asthma symptom diary as the number of occasions the reliever inhaler was used. An occasion is defined as 2 puffs for salbutamol or 1 inhalation for SYMBICORT.
  Standard deviation of total (daily) reliever medication use were presented for each patient and based on these summary statistics at treatment level were calculated.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Mean (Full Range); unit: Number of Occasions
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Number of Occasions | 0.75 [0.00 to 1.47] | 1.16 [0.31 to 2.75]

4. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Morning and Evening)
Description: FEV1 was measured by the patient using a spirometry sensor (Spirobank Smart™). Standard deviation of daily measurement of FEV1 were presented for each patient and based on these summary statistics at treatment level were calculated.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Mean (Full Range); unit: Liter (L)
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Liter (L)
  Morning | 0.169 [0.078 to 0.386] | 0.188 [0.089 to 0.576]
  Evening | 0.165 [0.079 to 0.361] | 0.197 [0.087 to 0.722]

5. Primary Outcome: Peak Expiratory Flow (PEF) (Morning and Evening)
Description: PEF was measured by the patient using a spirometry sensor (Spirobank Smart™). Standard deviation of daily measurement of PEF were presented for each patient and based on these summary statistics at treatment level were calculated.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Mean (Full Range); unit: Liter/minute (L/minute)
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Liter/minute (L/minute)
  Morning | 30.92 [16.20 to 59.51] | 36.28 [19.89 to 73.16]
  Evening | 30.17 [18.19 to 56.81] | 35.61 [22.86 to 79.42]

6. Secondary Outcome: Number of Patients With Secondary Objective Events
Description: The number of patients with inflammatory, asthma symptoms, lung function, and reliever use profile surrounding an event were assessed. Events of interest were Severe exacerbation (SevEx), composite surrogate endpoint for severe exacerbations of asthma (CompEx), and a single day (in 24 hours) with 6 or more occasions of reliever medication use.
  CompEx is an extended definition of asthma exacerbations combining diary-based event with traditionally defined severe exacerbations.
  Severe exacerbation are the events leading to one or more of the following; ≥ 3 days of oral corticosteroids (or one depot intramuscular injection of a glucocorticosteroid), an urgent care or emergency room visit that results in systemic corticosteroids, or an inpatient hospitalisation due to asthma.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Participants
  SevEx events | 2 | 7
  CompEx events | 4 | 12
  A single day (in 24 hours) with 6 or more occasions of reliever medication use | 3 | 9

7. Secondary Outcome: Number of Secondary Objective Events
Description: The inflammatory, asthma symptoms, lung function, and reliever use profile surrounding an event were assessed. Events of interest were Severe exacerbation (SevEx), composite surrogate endpoint for severe exacerbations of asthma (CompEx), and a single day (in 24 hours) with 6 or more occasions of reliever medication use.
  CompEx is an extended definition of asthma exacerbations combining diary-based event with traditionally defined severe exacerbations.
  Severe exacerbation are the events leading to one or more of the following; ≥ 3 days of oral corticosteroids (or one depot intramuscular injection of a glucocorticosteroid), an urgent care or emergency room visit that results in systemic corticosteroids, or an inpatient hospitalisation due to asthma.
Time Frame: From Day 1 to Day 169 (Treatment period)
Population: as for outcome 1
Measure: Number; unit: Number of events
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
Number analyzed (Participants) | 18 | 24
Number of events
  SevEx events | 2 | 8
  CompEx events | 8 | 15
  A single day (in 24 hours) with 6 or more occasions of reliever medication use | 3 | 18

ADVERSE EVENTS:
Time Frame: From Run-in period (Day -14 to -1) up to premature discontinuation visit and last Event Visit (Day 169)
Arm/Group | SYMBICORT as Maintenance and Reliever Treatment | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/24
Other Adverse Events (participants affected / at risk) | 0/18 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYMBICORT as Maintenance and Reliever Treatment (N=18) | SYMBICORT as Maintenance, Salbutamol as Reliever Treatment (N=24)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT03924635/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03924635/SAP_001.pdf